CLINICAL TRIAL: NCT06310408
Title: Comparison Between Nasal Mask vs Nasal Prong on Pain Response in Neonate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Besse Sarmila, dr, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0214022024
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Nasal Mask; Nasal Prong
Keywords: nasal mask, nasal prong, pain response

STUDY DESIGN:
Intervention Model Description: 1 group give nasal mask
  1 group give nasal prong
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal mask (Experimental): Give noninvasif respiratory support with interface nasal mask
  Interventions: Device: nasal mask
- nasal prong (Active Comparator): Give noninvasif respiratory support with interface nasal prong
  Interventions: Device: nasal prong

INTERVENTIONS:
Device: nasal mask — Give interface nasal mask
  Arms: nasal mask
Device: nasal prong — give interface nasal prong
  Arms: nasal prong

SUMMARY:
to determine the comparison of nasal masks and nasal prongs on the pain response of neonate

DETAILED DESCRIPTION:
To see the comparison of nasal masks and nasal prongs on the pain response of neonates, by measuring salivary cortisol levels before and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Newborn with espiratory distress and need noninvasive respiratory support

Exclusion Criteria:

* Syok, multiple congenital anomaly

Ages: 26 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
pain response | 20 weeks
  kortisol saliva level

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: i year